CLINICAL TRIAL: NCT03843034
Title: Endometrial Markers in Women With Autoimmune Diseases Receiving Assisted Reproduction
Brief Title: Endometrial Markers in Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, MD, PhD, Odense University Hospital
Other Study IDs: Lab.Reprod.Biol. - Odense.04
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Receptivity; Fertility; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Infertile women with autoimmune disease
  Interventions: Genetic: Measure endometrial markers
- Control group: Women from couples with severe male infertility
  Interventions: Genetic: Measure endometrial markers

INTERVENTIONS:
Genetic: Measure endometrial markers — Endometrial biopsies will be taken from participants in both groups

SUMMARY:
Autoimmune diseases cause a decreased endometrial receptivity during the implantation window, most likely changing the endometrial cytokines pattern due to dysregulation of the inflammatory processes.Therefore, endometrial cytokine profiles will be compared in women with autoimmune disease and normal, fertile women.

The collected endometrial tissue and blood samples will be examined for the cytokines profiling using commercially available ELISA kits.

The sample size was calculated choosing, as primary outcome, changes in endometrial LIF concentration between the disease and control Group, which is our main goal. Given a type I error of 5%, a maximum of 21 women are needed for each Group to reach the desired power of 80% to detect the least changes in concentrations.

ELIGIBILITY:
Inclusion Criteria:

Study group:

* Females with infertility combined with autoimmune disease and in fertility treatment.

Control group:

* Female from couples with severe male infertility and in fertility treatment.

Exclusion Criteria:

* Language problems to such an extent that the subjects do not understand the scope of the study.
* Abnormal follicle stimulating hormone (FSH),
* Abnormal antral follicles Count
* Genital infections
* Endometriosis
* Tubal occlusion
* Polycystic ovarian syndrome

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — It is a study on endometrial factors in female infertility
Study Population: Women with thyroid diseases, rheumatoid arthritis, inflammatory bowel diseases, multiple sclerosis, diabetes mellitus, and psoriasis will be included in the study Group (Age: 20-40 years old). Healthy women receiving assisted reproduction due to male infertility will be included in the control Group (Age: 20-40 years old).
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Endometrial cytokine LIF concentration (pg/ml) | February 18, 2019 - August 31, 2020
  The endometrial cytokine LIF profile in endometrial biopsies of women with autoimmune disease will be determined and compared to normal, fertile women (pg/mL)

SECONDARY OUTCOMES:
Blood concentration of cytokines such as LIF, IL6, TNFα TGFα (pg/ml) | February 18, 2019 - August 2020
  The blood cytokines concentration will be compared between the autoimmune diseases group and the control group. Moreover the cytokines concentration in blood and endometrial tissue will be compared.
endometrial concentration of cytokines such as, IL6, TNFα TGFα (pg/ml) | February 18, 2019 - August 2020
  The endometrial cytokines concentration will be compared between the autoimmune diseases group and the control group. Moreover the cytokines concentration in blood and endometrial tissue will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Andrology & Fertility Clinic, Department D, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No